CLINICAL TRIAL: NCT02839811
Title: Compact Biophotonic Platform for Drug Allergy Diagnosis
Brief Title: Medical Device for Drug Allergy Diagnosis
Acronym: COBIOPHAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9617
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Drug Hypersensitivity
Keywords: Betalactams; In vitro diagnosis
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- immediate hypersensitivity to BLC (Experimental): immediate hypersensitivity to BLC by In vitro diagnosis
  Interventions: Procedure: Immediate hypersensitivity to BLC

INTERVENTIONS:
Procedure: Immediate hypersensitivity to BLC — immediate hypersensitivity to BLC by In vitro diagnosis

SUMMARY:
The COBIOPHAD project targets the development of a highly sensitive, selective, and multiplexed diagnostic device to provide a quick and inexpensive in vitro test to address the most prevalent drug hypersensitivity to betalactams antibiotics, (BLCs). During a retrospective study, BLC structures involved in drug hypersensitivity will be identified from sera of allergic patients (versus controls) and coupled on the device.

A prospective study will be performed for the recruitment of samples corresponding to patients with known IgE hypersensitivity to BLCs based on results from allergy tests and clinical history. Controls will include: non-allergic individuals with known tolerance to betalactams. The samples will be used for the validation of the COBIOPHAD device in real settings.

ELIGIBILITY:
Inclusion Criteria:

- patients with known hypersensitivity to BLC (proven by means of in vivo tests) (cases)

Exclusion Criteria:

* patients with contraindications to BLC allergy work-up
* patient refusal to enter the study
* vulnerable patients according to French regulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the COBIOPHAD device in diagnosing immediate hypersensitivity to BLC | up to 1 hour
Specificity of the COBIOPHAD device in diagnosing immediate hypersensitivity to BLC | up to 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided